CLINICAL TRIAL: NCT06787781
Title: Metabolic and Clinical Effect of Alpha-lipoic Acid Administration in Schizophrenic Subjects Stabilized With Atypical Antipsychotics: A 12-week, Open-label, Uncontrolled Study
Brief Title: Metabolic and Clinical Effect of Alpha-lipoic Acid Administration in Schizophrenic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Fiammetta Iannuzzo, Principal investigator, University of Messina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: alphalipoic1
Record Dates: First submitted 2024-12-09; First posted 2025-01-22 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Evaluation; Cardiac Complications
Keywords: alphalipoic acid; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alpha Lipoid Acid (Experimental): Subject with schizophrenia administrated with ALA
  Interventions: Drug: Alpha Lipoic Acid

INTERVENTIONS:
Drug: Alpha Lipoic Acid — ALA was administrated in capsules at a xed oral daily dose of 600 mg for the entire duration of the study in addition to the atypical antipsychotic therapy.

SUMMARY:
The therapeutic use of ALA in schizophrenia has recently been investigated in human populations. A case series explored the effiacy of ALA as a novel agent to treat antipsychotic-induced obesity, at a dose of 1200 mg/d (range between 600 and 1800 mg/d); reporting the key effect to be a reduction in body weight and BMI after a 12-week treatment. In a pilot open-label trial, 100 mg/d of ALA was administrated as a general adjuvant to antipsychotics therapy, with no significant improvement in BMI, abdominal circumference, blood count, or liver enzymes. Finally, another study investigated the effects of 500 mg/d of ALA on plasma adiponectin levels, fasting glucose, and aspartate aminotransferase activity, with no significant effect on the metabolic parameters. Based on this background, ALA may be a potentially interesting therapeutic agent to improve the metabolic effects of atypical antipsychotics. The purpose of this study was to assess: (1) the efficacy of ALA on metabolic factors and (2) its safety and potential therapeutic effects in a sample of schizophrenic patients in stable therapy with atypical antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 criteria for schizophrenia,
* aged between 18 and 60 years old
* in stable atypical antipsychotic monotherapy (clozapine, olanzapine, quetiapine, or risperidone) for least 3 months.

Exclusion Criteria:

* treatment with more than one atypical antipsychotic, current treatment with insulin/oral hypoglycaemic/lipid-lowering agents
* significant concomitant medical pathologies
* organic brain disorders
* history of alcohol or substance dependence (excluding nicotine)
* dementia
* mental retardation
* pregnancy/breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iannuzzo F, Basile GA, Campolo D, Genovese G, Pandolfo G, Giunta L, Ruggeri D, Di Benedetto A, Bruno A. Metabolic and clinical effect of alpha-lipoic acid administration in schizophrenic subjects stabilized with atypical antipsychotics: A 12-week, open-label, uncontrolled study. Curr Res Pharmacol Drug Discov. 2022 Jun 28;3:100116. doi: 10.1016/j.crphar.2022.100116. eCollection 2022. PMID 35992380

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who met DSM-5 criteria for schizophrenia, aged between 18 and 60 years old in stable atypical antipsychotic monotherapy (clozapine, olanza- pine, quetiapine, or risperidone) for least 3 months.
Groups:
- AlphaLipoicAcid Group: Subject with schizophrenia administrated with ALA
Period: Overall Study
Arm/Group | AlphaLipoicAcid Group
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- AlphaLipoidAcid Group: Subject with schizophrenia administrated with ALA
Arm/Group | AlphaLipoidAcid Group
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.60 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 15
Body weight [Mean (Standard Deviation); unit: kg] | 95.80 (19.13)
Body massindex [Mean (Standard Deviation); unit: kg/m2] | 32.18 (5.99)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 137 (22.01)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 82 (15.49)
Qtc [Mean (Standard Deviation); unit: msec] | 422.80 (17.11)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 110.60 (57.01)
total cholesterol [Mean (Standard Deviation); unit: mg/dl] | 177.20 (39.62)
HDL [Mean (Standard Deviation); unit: mg/dl] | 38.8 (6.74)
LDL [Mean (Standard Deviation); unit: mg/dl] | 108.80 (33.93)
Glucose [Mean (Standard Deviation); unit: mg/dl] | 105.40 (14.05)
glycated haemoglobin [Mean (Standard Deviation); unit: percentage] | 5.20 (.53)
ALT [Mean (Standard Deviation); unit: U/L] | 28.80 (12.06)
AST [Mean (Standard Deviation); unit: U/L] | 23.20 (7.16)
gammaGT [Mean (Standard Deviation); unit: U/L] | 18.20 (7.06)
CPK [Mean (Standard Deviation); unit: U/L] | 203.40 (177.13)
creatinine [Mean (Standard Deviation); unit: mg/dl] | .86 (.17)
azotemia [Mean (Standard Deviation); unit: mg/dl] | 26.60 (4.14)
prolactinemia [Mean (Standard Deviation); unit: μUl/ml] | 389.76 (405.65)
Total score at the PANSS (Positive and Negative Syndrome Scale) [Mean (Standard Deviation); unit: units on a scale] — The PANSS (Positive and Negative Syndrome Scale) is a widely used tool for measuring the severity of schizophrenia symptoms. It assesses positive symptoms, negative symptoms, and general psychopathology in individuals with schizophrenia or related disorders.
  Cut off score of the scale: Total score (range 30-210); severity range: severity ranges:
  Mild symptoms: ~58-75 Moderate symptoms: ~75-95
  units on a scale | 72.80 (26.64)

OUTCOME MEASURES:

1. Primary Outcome: Assessing the Effect of ALA on the Blood Parameters: Lipid and Carbohydrate Framework
Description: Assessment of metabolic parameters: Total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), trigycerides, glucose
Time Frame: Assessed from enrollment to the end of treatment at 12 weeks, week 12 reported
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | AlphaLipoidAcid Group
Number analyzed (Participants) | 15
mg/dl
  total cholesterol | 180.60 (39.93)
  HDL | 37.60 (7.56)
  Glucose | 88.80 (12.56)
  Triglicerides | 132 (78.55)

2. Secondary Outcome: Total Score Changes Measured by Positive and Negative Schizophrenic Symptoms Scale (PANSS)
Description: The PANSS (Positive and Negative Syndrome Scale) is a widely used tool for measuring the severity of schizophrenia symptoms. It assesses positive symptoms, negative symptoms, and general psychopathology in individuals with schizophrenia or related disorders.
  Cut off score of the scale: Total score (range 30-210); severity range: severity ranges:
  Mild symptoms: ~58-75 Moderate symptoms: ~75-95 Marked symptoms: ~95-116 Severe symptoms: ~116+
Time Frame: Assessed from enrollment to the end of treatment at 12 weeks, week 12 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Alpha Lipoid Acid Group: Subject with schizophrenia administrated with ALA
  Alpha Lipoic Acid: ALA was administrated in capsules at a xed oral daily dose of 600 mg for the entire duration of the study in addition to the atypical antipsychotic therapy.
Arm/Group | Alpha Lipoid Acid Group
Number analyzed (Participants) | 15
score on a scale | 74.80 (34.21)

3. Other Pre Specified Outcome: Assessing the Effect of ALA on the Blood Parameters: Hepatic Framework
Description: alanineaminotransferase (ALT), aspartate aminotransferase (AST), gammaglutamyl transferase (γGT), creatine phosphokinase (CPK)
Time Frame: Assessed from enrollment to the end of treatment at 12 weeks, week 12 reported
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | AlphaLipoidAcid Group
Number analyzed (Participants) | 15
U/L
  ALT | 21.80 (9.76)
  AST | 17.80 (3.36)
  γGT | 15.60 (6.13)
  CPK | 84.20 (50.35)

4. Other Pre Specified Outcome: Assessing the Effect of ALA on the Blood Parameters: Renal Framework
Description: Creatinine, Azotemia
Time Frame: Assessed from enrollment to the end of treatment at 12 weeks, week 12 reported
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | AlphaLipoidAcid Group
Number analyzed (Participants) | 15
mg/dl
  creatinine | .88 (.13)
  azotemia | 30.80 (4.91)

5. Other Pre Specified Outcome: Assessing the Effect of ALA on the Blood Parameters: Electrocardiography
Description: QTc interval
Time Frame: Assessed from enrollment to the end of treatment at 12 weeks, week 12 reported
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | AlphaLipoidAcid Group
Number analyzed (Participants) | 15
msec | 408.80 (21.74)

6. Other Pre Specified Outcome: Assessing the Effect of ALA on BODY MASS INDEX
Description: body mass index
Time Frame: Assessed from enrollment to the end of treatment at 12 weeks, week 12 reported
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | AlphaLipoidAcid Group
Number analyzed (Participants) | 15
kg/m2 | 32.84 (5.63)

7. Other Pre Specified Outcome: Assessing the Effect of ALA on Blood Pressure
Description: systolic and diastolic blood pressure
Time Frame: Assessed from enrollment to the end of treatment at 12 weeks, week 12 reported
Measure: Mean (Standard Deviation); unit: mmg Hg
Arm/Group | AlphaLipoidAcid Group
Number analyzed (Participants) | 15
mmg Hg
  systolic blood pressure | 128 (18.07)
  diastolic blood pressure | 84 (14.68)

8. Other Pre Specified Outcome: Assessing the Effect of ALA on Prolactinemia
Description: prolactinemia
Time Frame: Assessed from enrollment to the end of treatment at 12 weeks, week 12 reported
Measure: Mean (Standard Deviation); unit: μUl/ml
Arm/Group | AlphaLipoidAcid Group
Number analyzed (Participants) | 15
μUl/ml | 190.16 (196.75)

ADVERSE EVENTS:
Time Frame: From enrollment to the end of treatment at 12 weeks
Description: No patient presented neither adverse effects nor undesirable change in the safety parameters
Groups:
- Alpha Lipoic Acid: Subject with schizophrenia administrated with ALA
  Alpha Lipoic Acid: ALA was administrated in capsules at a xed oral daily dose of 600 mg for the entire duration of the study in addition to the atypical antipsychotic therapy.
Arm/Group | Alpha Lipoic Acid
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
The small sample size, the lack of a comparative treatment, and the uneven distribution between sexes. Additionally, the length of the study was relatively short and thus it was not possible to assess the long-term effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT06787781/Prot_SAP_000.pdf